CLINICAL TRIAL: NCT00823459
Title: Phase II Trial of RAD001 in Patients With Recurrent Low Grade Glioma
Brief Title: Everolimus in Treating Patients With Recurrent Low-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Susan Chang (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Susan Chang, MD, Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08109; NCI-2011-01701 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 08109 (Other: UCSF Medical Center-Mount Zion); NCT00831324 (obsolete NCT alias)
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Adult Diffuse Astrocytoma; Adult Mixed Glioma; Adult Oligodendroglioma; Adult Subependymal Giant Cell Astrocytoma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Astrocytoma; Glioma; Oligodendroglioma; Brain Neoplasms | interventions — Everolimus

ARMS (1):
- Single-Arm Everolimus (Experimental): Single-arm study with patients receiving Everolimus orally once daily dosing of 10 mg continuously from Day 1 of study until progression of disease or unacceptable toxicity. In addition archival tissue will be analysed for markers of P13K/mTOR pathway activation.
  Interventions: Drug: Everolimus; Other: Archival Tissue Analysis

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Other: Archival Tissue Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well everolimus works in treating patients with recurrent low-grade glioma. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To determine progression-free survival at 6 months associated with use of RAD001 (everolimus) in patients initially diagnosed with low-grade glioma who undergo biopsy or subtotal resection at the time of recurrence with pathologic evidence of recurrent low-grade glioma (LGG).

SECONDARY OBJECTIVES:

1. To further delineate the safety profile of RAD001 in patients with recurrent LGG.
2. To assess overall survival (OS) in patients treated with RAD001.
3. To assess the objective response rate (ORR) in patients treated with RAD001.
4. To assess the correlation of protein kinase B (PKB)/Akt and phosphatase and tensin homolog (PTEN) expression with response, progression status by 6 months, and OS in patients treated with RAD001.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a Karnofsky performance status of >= 60
* Patients must have a life expectancy > 8 weeks
* All patients must sign an informed consent document indicating that they are aware of the investigational nature of this study
* Patients must sign an authorization for the release of their protected health information
* Patients must have a magnetic resonance imaging (MRI) scan performed within 14 days prior to initial protocol treatment
* Patients must be registered in the University of California at San Francisco (UCSF) Neuro-Oncology database prior to treatment with study drug
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hb) > 9 g/dL
* Serum bilirubin =< 1.5 x upper limit of normal (ULN)
* International normalized ratio (INR) < 1.5 (anticoagulation is allowed if target INR =< 1.5 on a stable dose of warfarin or on a stable dose of low molecular weight [LMW] heparin for > 2 weeks at the time of registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN
* Serum creatinine =< 1.5 x ULN
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND fasting triglycerides =< 2.5 x ULN; NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Patients must have histologically proven intracranial low-grade glioma at initial diagnosis; low-grade gliomas include: astrocytoma, oligodendroglioma and mixed oligoastrocytoma; pilocytic astrocytomas are excluded
* Patients must have unequivocal evidence for tumor recurrence or progression by histology as determined by review of pathology by an attending neuro-pathologist at UCSF
* If most recent histology shows progression to high grade glioma, patients must have had prior radiotherapy in order to be eligible
* Paraffin-embedded sections of tissue acquired from surgery at the time of suspected recurrence must be available for analysis
* Patients must have evidence for tumor recurrence or progression by MRI as determined by radiographic review of images by an attending neuro-oncologist or neuro-radiologist at UCSF
* If the steroid dose is increased between the date of the MRI and registration on the trial, a new baseline MRI is required; this MRI must be performed after >= 5 days on a stable dose of steroids
* An MRI must be used throughout the period of protocol treatment for tumor measurement
* Patients must have evaluable disease
* Patients may have had treatment (including radiotherapy) for any number of relapses prior to this recurrence
* Patients must be at least 4 weeks from the completion of any radiation therapy
* Patients must be less than 4 months from the surgical procedure for this recurrence
* Patients must have recovered from the toxic effects of prior therapy:

  * 4 weeks from any investigational agent
  * 4 weeks from prior cytotoxic therapy (except 6 weeks from nitrosoureas, 3 weeks from procarbazine, 3 weeks from vincristine)
  * 3 weeks for non-cytotoxic or biologic agents e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, tarceva, etc; note a 3-week washout is required for prior treatment with bevacizumab

Exclusion Criteria:

* Patients who have not recovered from the side effects of a major surgery or significant traumatic injury or patients that may require major surgery during the course of the study
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent; topical or inhaled corticosteroids, and treatment with low dose Decadron (=< 3 mg daily) are allowed
* Other than surgery, patients may not have therapy for this recurrence (including radiation); supportive care such as steroids or anti-epileptics does not constitute treatment of recurrence
* Patients must not have any significant medical illnesses that in the investigator?s opinion cannot be adequately controlled with appropriate therapy or would compromise the patient?s ability to tolerate this therapy
* Patients with a history of any other cancer (except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period; close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus; examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Gu?rin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* Uncontrolled brain or all leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York heart Association Class III or IV
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * Severely impaired lung function
  * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN (Note: Optimal glycemic control should be achieved before starting trial therapy)
  * Active (acute or chronic) or uncontrolled severe infections
  * Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C)
* A Hepatitis B/C blood test must be done at screening for all patients; patients who test positive for Hepatitis C antibodies and the Hepatitis B antigen are ineligible
* A known history of human immunodeficiency virus (HIV) seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Impaired lung function: O2 saturation 88% or less at rest on room air by pulse oximetry; if O2 saturation is =< 88% at rest, further pulmonary function tests (PFTs) should be ordered to confirm normal pulmonary function and eligibility
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods; adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug, by both sexes (women of childbearing potential [WOCBP] must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001)
* Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients who have received prior treatment with an mammalian target of rapamycin (mTOR) inhibitor (e.g., sirolimus, temsirolimus, everolimus)
* Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (e.g., sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-01-23 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Chang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Daily Intervention With RAD001: Single arm study: RAD001 will be administered orally as once daily dose of 10 mg (two 5 mg tablets) continuously from study day 1 until progression of disease or unacceptable toxicity. Patients will be instructed to take RAD001 in the morning, at the same time each day. RAD001 may be taken with or without food.
Period: Overall Study
Arm/Group | Daily Intervention With RAD001
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population is the same as the assigned participant flow.
Groups:
- Daily Intervention With RAD001: RAD001 will be administered orally as once daily dose of 10 mg (two 5 mg tablets) continuously from study day 1 until progression of disease or unacceptable toxicity. Patients will be instructed to take RAD001 in the morning, at the same time each day. RAD001 may be taken with or without food.
Arm/Group | Daily Intervention With RAD001
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months.
Description: Number of patients alive without progressive disease at 6 months. Assessment of progression was defined by RANO as a 25% increase in the sum of all the products of measurable lesions, clear worsening of any evaluable disease or any new lesion
Time Frame: At 6 months after treatment start
Population: All patients treated with study drug
Measure: Count of Participants; unit: Participants
Groups:
- Daily Intervention With RAD001: RAD001 will be administered orally as once daily dose of 10 mg (two 5 mg tablets) continuously from study day 1 until progression of disease or unacceptable toxicity. Patients will be instructed to take RAD001 in the morning, at the same time each day. RAD001 may be taken with or without food.
  RAD001: RAD001 will be administered orally as once daily dose of 10 mg (two 5 mg tablets) continuously from study day 1 until progression of disease or unacceptable toxicity. Patients will be instructed to take RAD001 in the morning, at the same time each day. RAD001 may be taken with or without food.
Arm/Group | Daily Intervention With RAD001
Number analyzed (Participants) | 58
Participants
  Grade II: number analyzed (Participants) | 47
  Grade II | 39
  Grade III/IV: number analyzed (Participants) | 11
  Grade III/IV | 6

2. Secondary Outcome: RAD001 Safety Profile in Patients With Recurrent LLG
Description: Grade 4-5 treatment related adverse events as defined by CTCAE 3.0
Time Frame: 13 months
Population: All patients treated from the time of registration until discontinuation of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Intervention With RAD001
Number analyzed (Participants) | 58
Participants | 0

3. Secondary Outcome: Objective Response Rate (ORR) in Patients Treated With RAD001.
Description: Objective response is defined as complete or partial response as defined by RANO criteria as determined by MRI and steroid requirement. Complete response was defined by disappearance of all measurable disease with minimal or no steroids; a partial response was defined as 50% in sum of all products in perpendicular diameters of all measurable lesions with no new lesions on stable or decreasing steroids.
Time Frame: 12 months
Population: All patients who were treated with study drug
Measure: Number; unit: participants
Arm/Group | Daily Intervention With RAD001
Number analyzed (Participants) | 58
participants | 0

4. Secondary Outcome: Overall Survival (OS) in Patients Treated With RAD001.
Description: Number of years from the day the patient started treatment until the date of death, an average of 5 years.
Time Frame: Time from registration till death, an average of 5 years
Population: All patients in study
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Daily Intervention With RAD001
Number analyzed (Participants) | 58
years | 5.2 [4 to NA] — Upper limit of confidence interval not reached due to insufficient number of patients with events

5. Secondary Outcome: To Assess the Correlation of Activation of the PI3K/mTOR Pathway With Survival
Description: Survival of patients with p-S6 staining of >19% (activated pathway)
Time Frame: 5 years
Population: Patients for which the molecular marker PI3K pathway activation was available
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Daily Intervention With RAD001
Number analyzed (Participants) | 50
years | 3.9 [3.4 to NA] — Upper bound not reached

ADVERSE EVENTS:
Time Frame: Time of study start with first day of study dosing until patient is removed from protocol treatment up to 12 months of therapy
Arm/Group | Daily Intervention With RAD001
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 6/58
Other Adverse Events (participants affected / at risk) | 18/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Intervention With RAD001 (N=58)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Pneumonitis/pulmonary infiltrates
Seizure (Nervous system disorders) | 2 (2) — Seizure
Fever (General disorders) | 1 (1) — Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)
Pain (Nervous system disorders) | 1 (1) — Pain-Head/headache
Infection (Infections and infestations) | 1 (1) — Infection with normal ANC or Grade 1 or 2 neutrophils - Meninges (meningitis)
Renal/Genitourinary (Renal and urinary disorders) | 1 (1) — Malilgnancy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Intervention With RAD001 (N=58)
Renal/Genitourinary (Renal and urinary disorders) | 1 (1) — Renal/Genitourinary malignancy, Urinary frequency/urgency
Diarrhea (Gastrointestinal disorders) | 14 (33)
Nausea (Gastrointestinal disorders) | 7 (8)
constipation (Gastrointestinal disorders) | 4 (4)
vomiting (Gastrointestinal disorders) | 2 (2)
mucositis/stomatitis (Gastrointestinal disorders) | 3 (9) — Oral cavity
mucosititis/stomatitis (Gastrointestinal disorders) | 2 (2) — Anus
Flatulence (Gastrointestinal disorders) | 1 (1)
seizure (Nervous system disorders) | 5 (6)
ataxia (Nervous system disorders) | 2 (2)
Dizzness (Nervous system disorders) | 2 (2)
neuropathy (Nervous system disorders) | 2 (2) — Motor
mood alteration (Nervous system disorders) | 1 (1) — Agitation
Mood Alteration (Nervous system disorders) | 1 (1) — Depression
Neuropathy (Nervous system disorders) | 1 (1) — Sensory
Speech Impairment (Nervous system disorders) | 1 (1) — dysphasia or aphasia
Syncope (Nervous system disorders) | 1 (1) — Fainting
Pain (Nervous system disorders) | 6 (12) — Headache
Pain (Gastrointestinal disorders) | 1 (1) — Abdominal NOS
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Back
Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Chest/Thorax
Infection (Infections and infestations) | 1 (1) — with Grade III or IV neurtophils (ANC < 1.0x 10e9/L) - Lung
Infection (Infections and infestations) | 1 (1) — With normal ANC or Grade 1 or 2 neurtrophils - meninges (meningitis)
Fatigue (General disorders) | 5 (9)
insomnia (General disorders) | 2 (3)
Fever (General disorders) | 1 (1) — In absence of neutropenia,where neutropenia is defined as ANC < 1.0 x 10e9/L
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — desquamation
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — acne/acneiform
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Generalized
Musculoskeletal/soft Tissue (Musculoskeletal and connective tissue disorders) | 1 (1) — Other
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Shortness of breath
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) — Pulmonary Infiltrates
Blurred vision (Eye disorders) | 1 (1)
lymphopenia (Blood and lymphatic system disorders) | 3 (5)
Leukocytes (Blood and lymphatic system disorders) | 2 (12)
Platelets (Blood and lymphatic system disorders) | 2 (6)
Neutrophils (Blood and lymphatic system disorders) | 2 (3) — ANC
Increased ALT (Metabolism and nutrition disorders) | 2 (3)
hypertriglyceridemia (Metabolism and nutrition disorders) | 6 (16) — Triglyceride, serum-high
Hypophosephatemia (Metabolism and nutrition disorders) | 4 (4) — Phosphate, serum - low
Hypercholesteremia (Metabolism and nutrition disorders) | 3 (5) — Cholesterol, serum-high
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) — Glucose, Serum - high
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) — Potassium, serum - high
Hypernatremia (Metabolism and nutrition disorders) | 1 (4) — Sodium, serum - high
ALT (Metabolism and nutrition disorders) | 2 (3) — Serum glutamic pyruvic transaminase - serum high

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-03-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT00823459/Prot_SAP_000.pdf